CLINICAL TRIAL: NCT00696072
Title: Randomized Phase II Trial of Letrozole With or Without Dasatinib as First and Second-line Treatment for Hormone Receptor-positive, HER2-negative Post-menopausal Breast Cancer That is Unresectable, Locally Recurrent or Metastatic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: US Oncology Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-185; USOR 06-185
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Dasatinib; Drug: Letrozole
- A2 (Active Comparator)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 100 mg once daily, up to 2 years
  Other Names: Sprycel; BMS-354825
  Arms: A1
Drug: Letrozole — Tablets, Oral, 2.5 mg, once daily, up to 2 years
  Other Names: Femara

SUMMARY:
The purpose of this study is to find out what effect the combination of letrozole (brand name: Femara) and dasatinib (brand name: Sprycel) has on metastatic breast cancer compared to letrozole alone

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Has histologic or cytologic diagnosis of breast cancer; evidence of unresectable locally recurrent or metastatic disease
* Has measurable or evaluable-only disease
* Is female, ≥18 yrs of age, post menopausal or surgically sterile
* HER2 negative, HR+, ER+ and/or PgR+ breast cancer
* 0-1 prior chemotherapy regimen for metastatic disease.
* Prior adjuvant or neoadjuvant chemotherapy completed at least 1 month prior
* Prior tamoxifen therapy is allowed
* No AI therapy for >1 year without recurrence

Exclusion Criteria:

* Pregnant or breast feeding
* Prior hormonal therapy for metastatic or locally recurrent disease
* >1 chemotherapy regimen for metastatic disease
* Pleural or pericardial effusion
* Serious cardiac condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (27):
  - Northern Arizona Hematology & Oncology Associates, Sedona, Arizona
  - Arizona Oncology Associates D.B.A. Hematology Oncology, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Institute - New Hope, Hudson, Florida
  - Central Indiana Cancer Centers, Carmel, Indiana
  - New York Oncology Hematology, Pc, Troy, New York
  - Dayton Oncology And Hematology, Kettering, Ohio
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Northwest Cancer Specialists, Pc, Portland, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Texas Oncology-Central Austin Cancer Center, Austin, Texas
  - Texas Oncology, Bedord, Texas
  - Texas Cancer Center At Medical City, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - El Paso Cancer Treatment Ctr - East, El Paso, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology, Garland, Texas
  - Texas Oncology, Houston, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Cancer Care Centers Of South Texas, San Antonio, Texas
  - Texas Oncology Cancer Center - Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care And Research Center, Waco, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematology Associates Of Southwest Virginia, Inc., Salem, Virginia
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started October 2008 and completed June 2014; 23 participants chose to remain on active treatment after the study completed.
Pre-assignment Details: 120 participants were enrolled, randomized and treated.
Groups:
- Dasatinib Plus Letrozole: Dasatinib + Letrozole: Tablets, Oral, once daily, up to 2 years
  Dasatinib 100 mg + Letrozole 2.5 mg Tablets, once daily up to 2 years. If a participant experienced intolerable toxicity related to dasatinib, they had the option to crossover to letrozole arm.
- Letrozole: Participants received letrozole 2.5 mg tablets, once daily, up to 2 years. If the participant developed progressive disease while on the single agent, the participant had the option to add dasatinib to their treatment regimen.
Period: Overall Study
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Started | 57 | 63
Completed | 0 | 0
Not Completed | 57 | 63
Not completed — continuing active treatment | 10 | 13
Not completed — Adverse Event | 10 | 6
Not completed — Patient Request | 3 | 7
Not completed — Investigator Request | 1 | 4
Not completed — Sponsor Request | 0 | 1
Not completed — Disease Progression | 32 | 30
Not completed — Non-specified | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population
Groups:
- Dasatinib Plus Letrozole: Dasatinib + Letrozole: Tablets, Oral, once daily, up to 2 years
  Dasatinib 100 mg + Letrozole 2.5 mg
- Total: Total of all reporting groups
Arm/Group | Dasatinib Plus Letrozole | Letrozole | Total
Number analyzed (Participants) | 57 | 63 | 120
Age, Customized [Number; unit: participants]
  Less than 65 years | 33 | 34 | 67
  Greater than or equal to 65 years | 24 | 29 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 120
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 63 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Benefit (CBR) and Number of Participants With CBR Having a Disease Free Interval (DFI) Greater Than 2 Years - Evaluable Population
Description: CBR=participants with complete response (CR) + participants with partial response (PR) + participants with stable disease (SD) for a length of time greater than, equal to 6 months. CR= Disappearance of all target lesions. No new lesions. PR= At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. SD= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum LD since the treatment started. Physical examination,radiological assessment, and bone scans (if applicable) were used to assess outcome.
Time Frame: First dose of study drug to last dose plus 7 days, up to study completion (approximately 6 years)
Population: Evaluable Population was defined as all treated participants who met the protocol-specified efficacy analyses requirements and who received at least 1 dose of randomized study drug. Participants presented in the treatment arm to which they were originally randomized.
Measure: Number; unit: participants
Groups:
- Dasatinib Plus Letrozole: Dasatinib + Letrozole: Tablets, Oral, once daily, up to 2 years
  Dasatinib 100 mg + Letrozole 2.5 mg
  Patients on letrozole plus dasatinib received both drugs until progressive disease (PD) or intolerable toxicity. If the intolerable toxicity was determined to be related to dasatinib, dasatinib was discontinued and the patient continued on single-agent letrozole. Although drugs were taken daily, cycle length was 28-days
- Letrozole: Letrozole: Tablets, Oral, 2.5 mg, once daily, up to 2 years
  Patients on letrozole who developed progressive disease continued letrozole, and dasatinib was added to their treatment regimen. Although drugs were taken daily, cycle length was 28-days
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Number analyzed (Participants) | 56 | 61
participants
  CBR (CR+PR+SD) | 40 | 40
  CBR, DFI <= 2 Years | 20 | 20
  CBR, DFI > 2 Years | 20 | 20

2. Secondary Outcome: Number of Participants With Complete Response, Partial Response, Stable Disease, and Disease Progression
Description: CR= Disappearance of all target lesions. No new lesions. PR= At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. SD= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum LD since the treatment started. Progression (PD): At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: First dose of study drug to last dose plus 7 days, up to study completion (approximately 6 years)
Population: All treated participants who met the protocol-specified efficacy analyses requirements and who received at least 1 dose of study drug were analyzed. The participants are analyzed as per the treatment arm to which they were originally randomized.
Measure: Number; unit: participants
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Number analyzed (Participants) | 56 | 61
participants
  CR | 1 | 0
  PR | 12 | 15
  SD | 32 | 30
  SD >=6 months | 27 | 25
  PD | 7 | 16
  Not Evaluable | 4 | 0

3. Secondary Outcome: Median Progression Free Survival (PFS) - Intent to Treat (ITT) Population
Description: PFS was measured in months. Progression=At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Study initiated 2008 and completed 2014.
Time Frame: Day 1 to Study Completion (approximately 6 years)
Population: ITT population includes all participants enrolled in the study. The participants were analyzed as per the treatment arm to which they were originally randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Number analyzed (Participants) | 57 | 63
months | 20.1 [10.7 to 28.4] | 9.9 [7.4 to 19.8]

4. Secondary Outcome: Percentage of Participants Best Overall Response After Change From Letrozole to Letrozole Plus Dasatinib
Description: Participants in single-agent letrozole treatment arm who developed progressive disease, could continue letrozole, and add dasatinib to their treatment regimen. CBR=participants with CR + participants with partial response (PR) + participants with SD for a length of time ≥6 months divided by the total number of participants (%). CR= Disappearance of all target lesions. No new lesions. PR= At least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. SD= Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) taking as reference the smallest sum LD since the treatment started. PD=At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: First dose of study drug to last dose plus 7 days, up to study completion (approximately 6 years)
Population: Participants who changed their treatment regimen from single-agent letrozole to letrozole + dasatinib during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Crossed Over From Letrozole to Letrozole + Dasatinib: These participants were randomized to receive letrozole 2.5 mg PO once daily. After developing progressive disease they continued letrozole, and were permitted to add 100 mg PO once daily dasatinib to their treatment regimen.
Arm/Group | Crossed Over From Letrozole to Letrozole + Dasatinib
Number analyzed (Participants) | 35
percentage of participants
  Best Response of SD | 34.3 [19.1 to 52.2]
  Best Response of SD ≥6 months | 22.9 [10.4 to 40.1]
  Best Response of CBR | 22.9 [10.4 to 40.1]
  Best Response of PD | 20.0 [8.4 to 36.9]
  Best Response Not Available | 2.9 [0.1 to 14.9]
  Best Response Not Evaluable | 2.9 [0.1 to 14.9]
  Best Response Pending | 40.0 [23.9 to 57.9]

5. Secondary Outcome: Percentage of Participants With PFS At 6 Months and At 12 Months - ITT Population
Description: Progression=At least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. ITT population: from time of first enrollment to first PD for all ITT participants.
Time Frame: At 6 months and at 12 months
Population: ITT population=Includes all participants registered on the study. n= number at risk
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Number analyzed (Participants) | 57 | 63
percentage of participants
  6 Month (n=39, 39) | 77.2 [63.3 to 86.4] | 66.2 [53.0 to 76.5]
  12 Month (n=29, 20) | 64.6 [49.8 to 76.1] | 42.9 [29.77 to 55.5]

6. Secondary Outcome: Median Time to Treatment Failure (TTF) - ITT Population
Description: Time to TTF was measured in months. The number of participants with events (PD or off treatment due to any reason) was evaluated. The first PD was defined as the event for cross over participants in the single- agent letrozole treatment arm to add dasatinib to their regimen.
Time Frame: First dose of study drug to last dose plus 7 days, up to study completion (approximately 6 years)
Population: ITT population: All participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Number analyzed (Participants) | 57 | 63
Months | 10.2 [5.8 to 18.5] | 9.2 [5.5 to 11.1]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation, Serious Adverse Events (SAEs), and Deaths
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: First dose of study drug to last dose plus 30 days, up to study completion (approximately 6 years)
Population: All participants who received at least one dose of study drug were summarized. The participants were analyzed as per the treatment arm to which they were originally randomized.
Measure: Number; unit: participants
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Number analyzed (Participants) | 57 | 63
participants
  Deaths | 11 | 16
  SAEs | 14 | 2
  AEs Leading to Discontinuation | 10 | 6

ADVERSE EVENTS:
Time Frame: First dose of study drug to last dose plus 30 days
Description: Study initiated 2008 and completed 2014.
Arm/Group | Dasatinib Plus Letrozole | Letrozole
Serious Adverse Events (participants affected / at risk) | 14/57 | 2/63
Other Adverse Events (participants affected / at risk) | 56/57 | 57/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Plus Letrozole (N=57) | Letrozole (N=63)
Hypersensitivity Reaction (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Insufficiency (Cardiac disorders) | 0 | 1
Congestive Heart Failure (Cardiac disorders) | 0 | 1
Coronary Insufficiency (Cardiac disorders) | 1 | 0
Effusion Pericardial (Cardiac disorders) | 0 | 1
CVA (Blood and lymphatic system disorders) | 2 | 0
Cholelithiasis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 1 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Nausea and Vomiting (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Fever (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Meningitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Failure Liver (Metabolism and nutrition disorders) | 0 | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture Bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Body Numbness (Nervous system disorders) | 1 | 0
Discomfort Abdominal (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Mood Altered (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Disease Heart Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Effusion Pleural (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cerebral Infarction (Vascular disorders) | 1 | 0
Failure Heart (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Plus Letrozole (N=57) | Letrozole (N=63)
Abdominal Pain (Gastrointestinal disorders) | 5 | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 4 | 1
Allergy (Immune system disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
ALT Increased (Investigations) | 3 | 3
Anemia (Blood and lymphatic system disorders) | 17 | 8
Ankles Swelling (Musculoskeletal and connective tissue disorders) | 1 | 3
Anorexia (Gastrointestinal disorders) | 5 | 6
Anxiety (Nervous system disorders) | 6 | 8
Appetite Decreased (Gastrointestinal disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6
AST Increased (Investigations) | 3 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 14
Blisters (Skin and subcutaneous tissue disorders) | 3 | 0
Breath Shortness (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cellulitis (Infections and infestations) | 3 | 2
Chest Pain (General disorders) | 2 | 3
Chills (General disorders) | 3 | 2
Common cold (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 14 | 9
Coughing (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Creatinine Serum increased (Investigations) | 4 | 3
Depression (Nervous system disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 18 | 12
Dizziness (Nervous system disorders) | 11 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 3
Dryness Vaginal (Reproductive system and breast disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Gastroesophageal reflux (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 26 | 21
Stomatitis (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 15 | 10
Neutropenia (Blood and lymphatic system disorders) | 13 | 5
Effusion Pericardial (Cardiac disorders) | 3 | 1
Hypertension (Cardiac disorders) | 7 | 1
Fatigue (General disorders) | 29 | 27
Weight Loss (Metabolism and nutrition disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 16 | 9
Flash Hot (Endocrine disorders) | 3 | 1
Hot Flashes (Endocrine disorders) | 18 | 18
Fever (Infections and infestations) | 2 | 5
Infection (Infections and infestations) | 4 | 6
Edema (Blood and lymphatic system disorders) | 5 | 1
Edema Periorbital (Blood and lymphatic system disorders) | 4 | 1
Swelling (Blood and lymphatic system disorders) | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 11
Fluid Retention in Tissues (Musculoskeletal and connective tissue disorders) | 3 | 2
Fracture Bone (Musculoskeletal and connective tissue disorders) | 4 | 4
Joint Pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain Flank (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain Knee (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain Neck (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain Pelvic (Musculoskeletal and connective tissue disorders) | 0 | 3
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 15 | 11
Insomnia (Nervous system disorders) | 10 | 8
Neuropathy (Nervous system disorders) | 4 | 2
Neuropathy Peripheral (Nervous system disorders) | 2 | 3
Taste Alteration (Nervous system disorders) | 4 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Effusion Pleural (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Infection Respiratory (Infections and infestations) | 5 | 1
Infection Upper Respiratory (Infections and infestations) | 6 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2
Urinary Tract Infection (Infections and infestations) | 7 | 5
Flu-like Symptoms (General disorders) | 0 | 3
Pain (General disorders) | 19 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.